CLINICAL TRIAL: NCT04697212
Title: Improving Communication and Healthcare Outcomes for Patients With Communication Disabilities: The INTERACT Trial
Brief Title: Improving Communication and Healthcare Outcomes for Patients With Communication Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Mayo Clinic (Other); University of Illinois at Chicago (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-3148
Record Dates: First submitted 2020-12-30; First posted 2021-01-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Communication Disabilities
Keywords: Patient-provider communication; Communication strategies; Healthcare outcomes
MeSH Terms: conditions — Communication Disorders | interventions — Patient Care Team

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare team- + patient-directed intervention (Experimental): Team education and patient tool
  Interventions: Behavioral: Healthcare team- + patient-directed intervention; Behavioral: Healthcare team-directed intervention
- Healthcare team-directed intervention (Active Comparator): Team education
  Interventions: Behavioral: Healthcare team-directed intervention

INTERVENTIONS:
Behavioral: Healthcare team- + patient-directed intervention — Participants will experience a clinical encounter with a healthcare team that has received training on evidence-based communication strategies for patients with communication disabilities, and will also complete a "patient prompt" list that elicits strategies that they prefer the healthcare team to use during their visit.
  Arms: Healthcare team- + patient-directed intervention
Behavioral: Healthcare team-directed intervention — Participants will experience a clinical encounter with a healthcare team that has received training on evidence-based communication strategies for patients with communication disabilities.

SUMMARY:
In the United States, 14% of all adults report a speech, language, voice, and/or hearing disability (collectively known as communication disabilities, CD). Patients with CD, experience inequities in receipt of and access to high-quality healthcare services, including primary care. Poor patient-provider communication is a significant contributor to these disparities. When healthcare providers use evidence-based communication strategies, patients with CD have improved communication outcomes and satisfaction. Unfortunately, providers rarely use the strategies in practice. The objective of this study is to compare the effectiveness and implementation of two interventions to increase primary care providers' use of communication strategies, improving the quality of their communication with patients with CD.

Using a stepped-wedge study design and guided by the RE-AIM framework, we will compare a healthcare team-directed intervention (training) to a healthcare team-directed intervention + patient-directed intervention (patient-prompt list). In the healthcare team-directed intervention, the team will receive training on evidence-based communication strategies for patients with CD. In the patient-directed intervention, patients with CD will complete a "patient prompt" list that elicits strategies that they prefer the healthcare team to use during their visit.

The primary aim of the study is to compare the effectiveness of the interventions on patient-reported experience in primary care practices across 4 healthcare systems using a stepped-wedge randomized controlled trial.

Hypothesis 1: Patients with CD will report a higher quality of health, more positive experience, and greater self-efficacy when they use the patient-directed tool (intervention A+B) as compared to patients with CD in the healthcare team education-only phase (intervention A).

Hypothesis 2. Providers will use more patient-centered communication and strategies with the patient-directed intervention.

The second aim is to examine the adoption, implementation, and short-term sustainability of the interventions.

DETAILED DESCRIPTION:
About 40 million people have a communication disability (CD), which includes hearing, speech, language, and voice disabilities. Compared to non-disabled patients, patients with CD are more likely to have a greater number of chronic conditions, and have higher rates of asthma, hypertension, emphysema, cardiovascular disease, diabetes and arthritis. Approximately one third of people with CD report the quality of their health as fair/poor as compared to only 11% of patients without CD. Patients with CD are 2-4 times more likely to report difficulty finding a provider than those without CD. When they do access care, they report that the quality of care and communication they receive is low.

Communication strategies that patients with CD require may vary, and providers need to elicit and then adapt to patients' preferences for communication strategies. Provider education and patient-prompt tool interventions have demonstrated effectiveness in general populations. Provider communication education significantly improves their patient-centered communication. Patient-prompt tools empower patients to identify topics and communication styles they prefer and then share this information with their healthcare provider. While provider education and patient-prompt tools have been proven effective, their effectiveness has not been compared in the primary care setting for patients with CD. Therefore, the aim of this study is to adapt these two types of interventions for patients with CD in the primary care setting and then compare their effectiveness at improving patient-reported health related quality of life and experience with care.

In this study we will conduct a stepped-wedge randomized control trial design. The study will take place at 4 sites that have unique contributions that will add to the generalizability and dissemination of the results. They are diverse in their geographic location, include academic and community clinics, represent urban and suburban locations, and include racially and ethnically diverse patients. Eight clinics, 2 at each site, will be part of the trial.

All participating clinic sites will receive the healthcare team-directed intervention (intervention A) and then will be randomized as to when they begin implementing the patient-directed tool (intervention B). The A versus A+B study design ensures all participating healthcare team members receive the training, as national policies require healthcare team members receive training on effective communication with patients with CD. We will randomize at the clinic-level cluster to eliminate spillover intervention effects amongst providers within the same clinic.

Participating healthcare team members will all receive the healthcare team-directed intervention (a general overview training about communication disabilities and communication strategies that can be used with patients) during the month preceding trial roll-out. Clinics will be randomized as to when they begin implementing the patient-directed tool, with a new clinic beginning every two months. One month prior to implementation, the healthcare team members will receive a booster education training, be introduced to the patient-directed tool, and alerted that they will be handed the completed tool by patients with CD during the patients' clinical encounters.

To measure patient and provider perceptions, both groups will complete a survey after the clinical encounter. A subset of encounters will be videotaped, and content analysis will document providers' use of patient-centered strategies and any adaptations made to the intervention strategies. Chart review will document patients' healthcare utilization over time. To understand providers' experiences with both interventions and perceptions of feasibility, healthcare team members will participate in qualitative focus groups and interviews at 3 time points.

The outcomes from this study may help create patient and provider training and tools that, if proven successful, could be disseminated to other healthcare arenas to improve patient-provider communication and ultimately improved health outcomes for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants: Individuals with a communication disability who receive care at participating study sites
* Healthcare team participants: Healthcare staff and providers at participating study sites

Exclusion Criteria:

* Patient participants: Individuals without a communication disability
* Healthcare team participants: Individuals who do not work at participating study sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health-Related Quality of Life | 1 week, 6 months
  One week following their clinical encounter, patients will complete the PROMIS Global Health measure, which includes 10 items that measure Health-Related Quality of Life. The measure includes items that ask the patient to rate their pain, fatigue and emotional wellbeing for the past 7 days. We will ask these questions again 6 months after the clinical encounter.
Patient Experience with the Clinical Visit | Baseline
  Following their clinical encounter, patients will complete 2 subscales of the Patients' Perceptions of Quality of Care (PPQC) survey; Providers' Bedside Manner and Providers' work. Both subscales include questions about the quality of communication with their provider during their appointment. The PPQC has been demonstrated to detect differences in experience between patients with and without disabilities in the primary care setting.

SECONDARY OUTCOMES:
Provider Use of Communication Strategies | Baseline
  Providers' use of patient-centered communication and strategies will be measured through a content analysis of video-recorded clinical encounters of a subset of patients. The recorded video will be analyzed using the Roter Interaction Analysis System (RIAS), which is a coding system that will yield the ratio of the degree of patient-centered communication in the clinical encounter.
Patient Self-Efficacy for Management of Chronic Conditions | 1 week
  One week following the clinical encounter, patients will complete the PROMIS Global Health measure, which includes 8 items that measure Self-Efficacy for Management of Chronic Conditions. The measure includes items that ask about patients' self-efficacy for managing medications, treatments, and symptoms.
Provider Satisfaction with Quality of Interaction | Baseline
  Providers' perceptions of the communication will be measured using the Physician Satisfaction with Primary Care Office Visits survey, which has been used concurrently with the RIAS coding system to assess providers' perspectives of communication with diverse populations. The survey includes 20 items on a Likert scale.

OTHER OUTCOMES:
Patient Hospital Admissions | 6 months
  Electronic Health Record data will identify the number of hospital admissions among participating patients.
Patient Emergency Department (ED) Use | 6 months
  Electronic Health Record data will identify the frequency of ED use among participating patients.

CONTACTS AND LOCATIONS:
Overall Officials: Megan A Morris, PhD, MPH, Principal Investigator — New York University
Locations (5):
- United States (5):
  - Denver Health, Denver, Colorado
  - UCHealth Primary Care - Lone Tree, Lone Tree, Colorado
  - University of Illinois Chicago, Chicago, Illinois
  - Michigan Medicine, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD at this time.